CLINICAL TRIAL: NCT05362630
Title: Infliximab Efficacy in Relation to Therapeutic Drug Monitoring and Serum Tumor Necrosis Factor (TNF)α Levels in Pediatric HSCT Recipients With Acute Graft-versus-host Disease: a Prospective Observational Study
Brief Title: Infliximab Efficacy, TDM and Serum TNFα Levels in Pediatric HSCT Recipients With aGVHD: Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonello Di Paolo, M.D., Ph.D., Associate Professor of Pharmacology, University of Pisa
Other Study IDs: 441/2022
Record Dates: First submitted 2022-04-30; First posted 2022-05-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Graft Versus Host Disease, Acute; Hematopoietic Stem Cell Transplantation
Keywords: Graft-Versus-Host Disease; Hemopoietic Stem Cell Transplant; Infliximab; Therapeutic Drug Monitoring; Clinical response; Population Pharmacokinetic Analysis
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples to quantitate TNFalpha and infliximab concentrations
Oversight: Data Monitoring Committee: No

SUMMARY:
In children receiving a hematopoietic stem cell transplant (HSCT), blood levels of TNFalpha (an inflammatory cytokine) at the onset of the acute GVHD (graft-versus-host disease) could be correlated with the severity of the disease. The hypothesis is that the highest infliximab (a biologic drug against TNFalpha) could be associated with a significant reduction in TNFa levels and, subsequently, with a faster remission of the symptoms and prevention of disease progression. Moreover, a rapid drop of infliximab serum concentration, documented by therapeutic drug monitoring (TDM), could be related to the active phase of GVHD and higher production of TNFalpha. Therefore, the study is aimed at investigating whether the drop in infliximab plasma concentrations could be associated with clinical response and production of TNFalpha.

HSCT children receiving infliximab to control GVHD are enrolled. Blood samples will be collected during treatment and they serve to measure drug and TNFalpha concentrations. Drug levels are analyzed by a population pharmacokinetic modeling and results are compared with plasma concentrations of TNFalfa and clinical response.

DETAILED DESCRIPTION:
Despite significant progress in overall survival and event-free survival in Pediatric Hematopoietic Stem Cell Transplant (HSCT), therapeutic options for graft-versus-host disease (GVHD) control remain limited, particularly in steroid-refractory patients. Several strategies have been proposed in the last 20 years but so far the results have been mixed and inconclusive, complicated by the small population afflicted, inconsistent treatment schedules, diverse disease classifications, and diagnosis methods. The number of studies concerning pediatric patients is even smaller.

First-line therapy for acute GVHD is steroid treatment that achieves partial or complete remission of the disease in a variable percentage (40-60%) of cases, depending mainly on the severity of GVHD and number of organ involvement. Notably, hepatic and gastrointestinal GVHD is particularly refractory to steroid treatment.

For second-line therapy, there is no standardized strategy with a great variety of immunosuppressive treatments without a real superiority of a drug in comparison to another.

Steroid refractory acute GVHD is therefore one of the most important challenges in the HSCT field. One of the more promising routes, based on published data and clinical experience, is the off-label use of Infliximab, an anti-Tumor Necrosis Factor (TNF)alpha drug (already approved for many rheumatological and autoimmune diseases) administered as a second-line treatment in patients with steroid-refractory acute GVHD at the standardized dosage of 10 mg/kg, although, to our knowledge, no substantial evidence has been published to validate this subscription. The biological pattern that could explain the susceptibly of GVHD to infliximab treatment could lie in the physiopathology of acute gastrointestinal GVHD that may resemble ulcerative rectocolitis. In this case, relation to Therapeutic Drug Monitoring (TDM) and TNFalpha levels could be critical in monitoring the efficacy of the drug and the need for further doses.

Published data, scarce as it may be, and clinical experience showed that infliximab may be able to further control symptoms and inflammatory response in a promising percentage of treated patients, although some have no benefit from the treatment.

Therefore, the study is aimed at evaluating the role of TNFalpha concentration in acute GVHD, the fluctuation of its plasma levels, and the clinical response of GVHD to infliximab treatment in steroid-refractory pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HSCT recipient;
* Onset of clinical signs of acute skin, gastrointestinal or hepatic GVHD according to the Glucksberg classification;
* At least five days of steroid treatment (minimum 1 mg/kg of methylprednisone or equivalent) for systemic aGVHD without clinical or laboratory signs of response or no steroid treatment for onset of grade I-II hepatic/gastroesophageal/intestinal isolated aGVHD;
* Patients who consent for the off-label use of infliximab and data processing for research purposes based on the institutional model GECO;
* At least one dose of infliximab received during aGVHD management;
* Minimum follow-up after infliximab administration: 6 months

Exclusion Criteria:

* Follow up < 6 months.
* Active fungal or bacterial infection with life-threatening clinical condition (shock or respiratory distress that needs mechanical ventilation)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (0-18 years old) who undergo a HSCT and subsequently, develop an acute GVHD and receive infliximab
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation between TNFalpha and infliximab plasma concentrations at day +56 of treatment | Day 56 after the start of infliximab administration
  Correlation analysis between TNFalpha and infliximab plasma concentrations at day +56 of treatment

SECONDARY OUTCOMES:
Correlation between TNFalpha and infliximab plasma concentrations at day +7 of treatment | Day +7 after the start of infliximab administration
  Correlation analysis between TNFalpha plasma concentrations at day +7 of treatment
Relationship between baseline TNFalpha plasma concentration and aGVHD overall severity | From day -7 up to day -1 from the start of infliximab administration
  Correlation analysis between TNFalpha plasma concentrations and the severity of aGVHD
Clinical response to infliximab | Day +56 of treatment
  Percentage of patients who achieve Complete Response (CR), Partial Response (PR), Non-Response (NR) to infliximab treatment for acute GVHD
Infliximab plasma concentrations according to clinical response | From day +7 up to day +56 of treatment
  Values of plasma concentrations of infliximab according to complete response, partial response and no-response (CR, PR, NR, respectively)
Percentage of transplant-related deaths and infections during follow-up | From +6 months up to +1 year after treatment
  Percentage of transplant-related mortality (TRM), viral reactivation (EBV, CMV), bacterial and fungal infection during follow-up
Retreatment rate with infliximab after the first dose | From +90 days from treatment begin up to +1 year
  Percentage of patients who require a new treatment with infliximab after at least 3 months after the first course
Safety of drug treatment | From day +100 up to +1 year post-HSCT
  Percentage of patients who survive and free from bacterial and fungal infections after HSCT
Overall survival (OS) | From day +100, up to +1 year after HSCT
  OS after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Maximova, MD, Study Director — IRCCS Burlo Garofolo - Trieste, Italy
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maximova N, Nistico D, Riccio G, Maestro A, Barbi E, Faganel Kotnik B, Marcuzzi A, Rimondi E, Di Paolo A. Advantage of First-Line Therapeutic Drug Monitoring-Driven Use of Infliximab for Treating Acute Intestinal and Liver GVHD in Children: A Prospective, Single-Center Study. Cancers (Basel). 2023 Jul 13;15(14):3605. doi: 10.3390/cancers15143605. PMID 37509268